CLINICAL TRIAL: NCT06074640
Title: Effects of Post Isometric Relaxation With and Without Dry Needling in Triceps Surae With Chronic Heel Pain.
Brief Title: Effects of PIR With and Without Dry Needling on Heel Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0163Maham Khurshid
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Heel Pain Syndrome
Keywords: chronic heel pain; dry needling; post isometric relaxation; tricep surae; trigger points
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group 1(MET PIR with Dry needling) (Experimental): Participants of this group will be treated with a MET protocol, and a dry needling session for Calf muscles MTrPs. Home regimen of self stretches for Calf muscles and plantar fascia will be given to patients
  Interventions: Other: MET PIR with Dry Needling
- interventional group II (MET PIR without dry needling) (Experimental): participants will follow the same MET PIR exercises but without adjunct dry needling for Calf muscles. Home regimen of self stretches for Calf muscles and plantar fascia will be given to patients
  Interventions: Other: MET PIR without Dry Needling

INTERVENTIONS:
Other: MET PIR with Dry Needling — MET PIR Protocol: The subject will be asked to exert a small effort (20% of available strength) towards plantar flexion, against unyielding resistance, for 20 seconds. Once released, ankle will be dorsiflexed beyond the new range gained and stretched for up to 30 seconds. Rest period will be of 1 minute in between each repetition. (3 Repetitions, 1 Sets, 3 days per week, for 4 weeks consecutively.) MTrPs will be identified and located using flat or pincer palpation method in the Triceps Surae complex of the affected leg. The identified trigger points will be marked with a marker. Piston technique of dry needling is performed on the identified MTrPs in calf muscles. The self stretches of Plantar Fascia and Calf muscles will be demonstrated. The stretch position will be maintained for 20 sec, followed by 20 sec rest and then repeated for 3 minutes. All stretches will be performed twice daily by patients for 4 weeks time period (3 Reps, 2 sets/day, for 4 weeks)
  Arms: interventional group 1(MET PIR with Dry needling)
Other: MET PIR without Dry Needling — MET PIR Protocol: The subject will be asked to exert a small effort (20% of available strength) towards plantar flexion, against unyielding resistance, for 20 seconds. Once released, ankle will be dorsiflexed beyond the new range gained and stretched for up to 30 seconds. Rest period will be of 1 minute in between each repetition. (3 Repetitions, 1 Sets, 3 days per week, for 4 weeks consecutively.) The self stretches of Plantar Fascia and Calf muscles will be demonstrated. The stretch position will be maintained for 20 sec, followed by 20 sec rest and then repeated for 3 minutes. All stretches will be performed twice daily by patients for 4 weeks time period (3 Reps, 2 sets/day, for 4 weeks)
  Arms: interventional group II (MET PIR without dry needling)

SUMMARY:
The aim of this research will be to determine the effects of Post Isometric relaxation exercises with and without dry needling of triceps surae MTrPs on heel pain, ankle ROM and foot function in chronic heel pain patients. The sample size calculated for this study was 42. The subjects will be divided in two groups, 21 subjects in PIR with dry needling group and 21 in PIR without dry needling group. Study duration will be of 6 months. Sampling technique applied will be non probability convenience sampling technique. Only patients who are 20 - 40 years old, have NPRS score of heel pain above 3 and have MTrPs in any of the triceps surae muscle on initial inspection are included. Tools used in the study are Goniometer, NPRS scale and Foot function Index. Data will be analyzed through SPSS 23.

DETAILED DESCRIPTION:
A number of patients visit clinics with a common subjective complaint of heel pain, especially with advancing age. Chronic PHP is characterized by painful inferioromedial aspect of calcaeneum, tender to even palpation. Myofascial pain syndrome cause regional pain and its hallmark feature is the presence of trigger points in the affected muscles. Triggers points in triceps surae i.e. Gastro-soleus can generate symptoms in the vicinity or spill them over to heel, causing pain and restricted mobility. Manual therapy and acupuncture are tools to deactivate MTrPs whilst restoring the muscle to its normal length and full joint range of motion with exercises and stretches. Dry needling treats trigger points by disrupting the tender points; whereas Post isometric relaxation is a form of muscle energy technique that restores the stretch length of a shortened, hypertonic muscle thereby decreasing myofascial pain. The aim of current RCT will be to compare the effects of post isometric relaxation with and without dry needling for trigger points of triceps surae in chronic heel pain patients.

Former studies have been conducted to explore the effects of various conventional and complementary therapies for heel pain rehabilitation. These studies provide evidence for the effectiveness of Muscle energy techniques and dry needling, as isolated treatments, in improving outcome measures for heel pain. Sufficient evidence also supports the efficacy of manual therapies with dry needling for neck pain, low back pain, knee or shoulder pain etc but is scarce for heel pain cases. Our study will apply multimodal approach by combining conventional stretching exercise and MET PIR with dry needling. Evidence of such a study published previously is almost negligible for heel pain rehab

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 40 yrs
* Both Genders (Males and Females)
* Clinical diagnosis of plantar heel pain in accordance with ICFDH
* Primary c/o unilateral heel pain on the inferomedial surface
* Pain elicited with first steps after waking
* Pain worsens on prolonged weight bearing or inactivity.
* Complaint of Heel Pain ≥ 6 month (Chronic)
* NPRS score of heel pain between scores above 3
* Ankle dorsiflexion less than 10° with extended knee or less than 20° with flexed knee.
* Presence of MTrPs in any of the triceps surae muscle (Gastrocnemius, soleus) on initial inspection

Exclusion Criteria:

* Patients with bilateral heel pain (may be systemic)
* Heel pain with absence of trigger points in Triceps surae complex.
* Participants diagnosed with serious causes of heel pain. (Ankle/foot fractures, Tumors etc)
* Secondary causes of heel pain(Congenital deformity, systemic inflammatory, vascular or neurological disorders etc)
* History of treatment for heel pain in the past 4 weeks
* Persons contraindicated for Acupuncture/Dry Needling

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Heel Pain | 4 weeks
  Heel pain scoring via NPRS Scale. This 11-point scale ranges from "0" interpreted as "No pain" to "10' interpreted as "worst imaginable pain" Change will be measured from baseline to 4 weeks.
Ankle Dorsiflexion ROM | 4 weeks
  Universal goniometer measurements of dorsiflexion range at Ankle. It has markings on its surface from 0° to 360° to measure ankle range of motion. Change will be measured from baseline to 4 weeks.

SECONDARY OUTCOMES:
Foot Function | 4 weeks
  Foot function index is used to assess foot function level. The FFI Questionnaire consists of 23 self-reported items divided into 3 subcategories on the basis of patient values: pain, disability and activity limitation. The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help), that best describes their foot over the past week. Change will be measured from baseline to 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Ashraf, TDPT, Principal Investigator — Riphah International University; Maham Khurshid, MS OMPT*, Principal Investigator — Riphah International University
Locations (1):
- Fatima Bashir Hospital, Ghakhar, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No